CLINICAL TRIAL: NCT01401101
Title: Improving PTSD Management in Primary Care
Brief Title: Violence and Stress Assessment (ViStA) Project to Improve Post Traumatic Stress Disorder Management in Primary Care
Acronym: ViStA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Clinical Directors Network (Network); Georgetown University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1R01MH082768 (NIH)
Record Dates: First submitted 2010-08-26; First posted 2011-07-25 (Estimated); Results first posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-07

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: mental health; PTSD; primary care; quality improvement; collaborative care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTSD Care Management (PCM) (Experimental): PCM has six intervention components: 1) patient education, 2) patient screening and written feedback of screening information to primary care clinicians, 3) clinician education on practice guidelines , 4) structured feedback between primary care and mental health clinicians, 5) continuity of patient care, and 6) a resource guide detailing available community services where the FQHC has established reciprocal referrals. All of the intervention components will be implemented through the CM, except for the clinician education component, which will combine onsite and online continuing medical education (CME)-accredited sessions.
  Interventions: Other: PCM
- Minimally Enhanced Usual Care (MEU) (Placebo Comparator): The MEU condition consists of only the clinician education and patient screening without written feedback.
  Interventions: Other: MEU

INTERVENTIONS:
Other: PCM — Care Manager (CM) intervention
  Arms: PTSD Care Management (PCM)
Other: MEU — The MEU condition consists of only the clinician education and patient screening without written feedback.
  Arms: Minimally Enhanced Usual Care (MEU)

SUMMARY:
The purpose of this study is to conduct a randomized trial of a Post Traumatic Stress Disorder (PTSD) Care Management (PCM) program to detect, treat, and improve PTSD treatment processes and outcomes in patients seeking primary care from FQHCs and evaluate its effectiveness on improving the processes and outcomes of care for PTSD.

DETAILED DESCRIPTION:
Post-traumatic Stress Disorder (PTSD) is a common problem seen in primary care but the identification and management of PTSD is not routine and would benefit from new approaches. Efforts must overcome patient-, clinician-, and system-level barriers, such as patients' fear of stigma, clinician's time constraints for dealing with psychological issues, gaps in clinician treatment knowledge, and difficulty arranging for referrals to mental health specialists.

Unlike mood disorders such as depression, little is known about improving care for PTSD in primary care settings. However, previous experience for treating depression, as well as existing guidelines for addressing PTSD in primary care, provide evidence that effective interventions exist and that multi-faceted interventions are more effective than a single-component approaches.

In this project, the RAND Corporation, Clinical Directors Network Inc., Georgetown University Department of Psychiatry, and University of Washington will implement and evaluate a randomized controlled trial (RCT) of a PTSD Care Management (PCM) intervention to detect, treat, and improve PTSD treatment processes and health outcomes in patients seeking primary care from Federally Qualified Health Centers (FQHCs) in Northeastern USA.

The three specific aims are to:

1. Evaluate the effectiveness of the PCM intervention compared to a minimally enhanced usual care (MEU) control in reducing PTSD and other mental health symptoms, and improving patients' health-related quality-of-life.
2. Assess the success of the PCM intervention implementation and,
3. Examine the direct costs of the PCM intervention compared to the TAU control treatment.

The PCM intervention was developed using principles of Community-Based Participatory Research (CPBR) methods in FQHCs that provide care to the underserved, and is tailored to the settings and populations we will study. This intervention is multi-faceted and includes components and strategies implemented through a Care Manager (CM) to overcome patient-, clinician-, and system-level barriers.

There are six PCM intervention components: 1) patient education, 2) patient screening and written feedback of screening information to primary care clinicians, 3) clinician education on practice guidelines , 4) structured feedback between primary care and mental health clinicians, 5) continuity of patient care, and 6) a resource guide detailing available community services where the FQHC has established reciprocal referrals. All of the intervention components will be implemented through the CM, except for the clinician education component, which will combine onsite and online continuing medical education (CME)-accredited sessions. The MEU condition will consist of only the clinician education and patient screening without written feedback.

Patients will be interviewed during a pre-screening stage to determine PTSD status. A total of 400 of the patients who screen positive will be randomly assigned to the PCM intervention or TAU.

Data will be collected from several sources. First, patients will be assessed at baseline, 6 and 12 months via interviews using validated instruments. Second, CMs will compile monthly aggregate data on patient management for patients assigned to the PCM program. Third, FQHC staff will be asked for their feedback about their experiences with implementing the program at the end of the study. The study team will use these data to estimate the direct costs of implementing the PCM program.

ELIGIBILITY:
Inclusion Criteria:

* Has PTSD
* Has a scheduled or walk-in appointment with a participating PCC
* Speaks English of Spanish
* Is between 18 and 65 years old
* Expects to receive care in the CHC during the next year

Exclusion Criteria:

* Acutely ill and cannot participate in a discussion
* Does not understand the information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2010-06; Primary Completion 2014-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Meredith, PhD, Principal Investigator — RAND
Locations (7):
- United States (7):
  - Metropolitan Family Health Center, Jersey City, New Jersey
  - Joseph P. Addabbo Health Centere, Far Rockaway, New York
  - Ryan NENA Health Center, New York, New York
  - Open Door Family Medical Center, Port Chester, New York
  - Morris Heights Health Center (Walton), The Bronx, New York
  - Community Health Care Network (Bronx Center), The Bronx, New York
  - Soundview Health Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
No data sharing plan was associated with this project at the time it was funded.

REFERENCES:
- [Background] Meredith LS, Eisenman DP, Green BL, Kaltman S, Wong EC, Han B, Cassells A, Tobin JN. Design of the Violence and Stress Assessment (ViStA) study: a randomized controlled trial of care management for PTSD among predominantly Latino patients in safety net health centers. Contemp Clin Trials. 2014 Jul;38(2):163-72. doi: 10.1016/j.cct.2014.04.005. Epub 2014 Apr 18. PMID 24747932
- [Background] Meredith LS, Eisenman DP, Han B, Green BL, Kaltman S, Wong EC, Sorbero M, Vaughan C, Cassells A, Zatzick D, Diaz C, Hickey S, Kurz JR, Tobin JN. Impact of Collaborative Care for Underserved Patients with PTSD in Primary Care: a Randomized Controlled Trial. J Gen Intern Med. 2016 May;31(5):509-17. doi: 10.1007/s11606-016-3588-3. Epub 2016 Feb 5. PMID 26850413

RESULTS

PARTICIPANT FLOW:
Groups:
- PTSD Care Management (PCM): There are six PCM intervention components: 1) patient education, 2) patient screening and written feedback of screening information to primary care clinicians, 3) clinician education on practice guidelines , 4) structured feedback between primary care and mental health clinicians, 5) continuity of patient care, and 6) a resource guide detailing available community services where the CHC has established reciprocal referrals. All of the intervention components will be implemented through the CM, except for the clinician education component, which will combine onsite and online continuing medical education (CME)-accredited sessions.
  quality improvement: Care Manager (CM) intervention
- Treatment-as-Usual (TAU): The TAU condition will consist of only the clinician education and patient screening without written feedback.
  Treatment-as-Usual: The TAU condition will consist of only the clinician education and patient screening without written feedback.
Period: Overall Study
Arm/Group | PTSD Care Management (PCM) | Treatment-as-Usual (TAU)
Started | 206 | 198
Completed | 184 | 171
Not Completed | 22 | 27

BASELINE CHARACTERISTICS:
Population: We randomized 206 patients to the PCM condition and 198 to the ECE conditions. However, only 355 patients of the 404 patients randomized completed the baseline survey, So, 49 patients have missing data in the evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | PTSD Care Management (PCM) | Treatment-as-Usual (TAU) | Total
Number analyzed (Participants) | 184 | 171 | 355
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.4) | 42.2 (12.0) | 42.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 136 | 286
  Male | 34 | 35 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 90 | 185
  Not Hispanic or Latino | 79 | 67 | 146
  Unknown or Not Reported | 10 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 95 | 88 | 183
  Asian | 64 | 60 | 124
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 7 | 21
  White | 0 | 1 | 1
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 184 | 171 | 355

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms
Description: Clinician-Administered PTSD Scale (CAPS) severity score: sum of ratings (from 0-4) for frequency and intensity across each of the 17 symptom items for a possible range of 0-136, where a higher score indicated higher severity.
Time Frame: 0 months (baseline)
Population: all patients who completed the assessment
Measure: Mean (95% Confidence Interval); unit: CAPS scores
Arm/Group | PTSD Care Management (PCM) | Treatment-as-Usual (TAU)
Number analyzed (Participants) | 184 | 171
CAPS scores | 71.1 [67.9 to 74.3] | 71.0 [67.9 to 74.2]
Statistical Analysis 1: Comparison: PTSD Care Management (PCM) vs Treatment-as-Usual (TAU); Intent-to-treat (ITT) analysis using the linear mixed-method model to estimate the difference between the PCM and TAU conditions; Test type: Superiority or Other; p = 0.97, Regression, Linear — Jointly modeled outcomes at the 3 waves by time, condition, and timeXcondition, to allow for different effects at 6 and 12 mos; controlled for interview mode (phone vs. in-person); used random effects to account for correlations wi/in site & patient

2. Primary Outcome: PTSD Symptoms
Description: same as baseline
Time Frame: 6 months
Population: Clinician-Administered PTSD Scale (CAPS) severity score: sum of ratings (from 0-4) for frequency and intensity across each of the 17 symptom items for a possible range of 0-136, where a higher score indicated higher severity.
Measure: Mean (95% Confidence Interval); unit: CAPS scores
Arm/Group | PTSD Care Management (PCM) | Treatment-as-Usual (TAU)
Number analyzed (Participants) | 184 | 171
CAPS scores | 47.8 [44.2 to 51.3] | 49.5 [46.4 to 52.6]
Statistical Analysis 1: Comparison: PTSD Care Management (PCM) vs Treatment-as-Usual (TAU); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.54, Regression, Linear

3. Primary Outcome: PTSD Symptoms
Description: same as baseline and 6 months
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: CAPS scores
Arm/Group | PTSD Care Management (PCM) | Treatment-as-Usual (TAU)
Number analyzed (Participants) | 184 | 171
CAPS scores | 46.9 [42.8 to 50.9] | 44.2 [41.2 to 47.1]
Statistical Analysis 1: Comparison: PTSD Care Management (PCM) vs Treatment-as-Usual (TAU); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.33, Regression, Linear — Jointly modeled outcomes at the 3 waves by time, condition, and timeXcondition, to allow for different effects at 6 and 12 mos; controlled for interview mode (phone vs. in-person); using random effects to control for correlations w/in site & patient

ADVERSE EVENTS:
Description: This study only monitored suicidal ideation as a non-serious adverse event. we also monitored suicide as a serious adverse events.
Groups:
- PTSD Care Management (PCM): There are six PCM intervention components: 1) patient education, 2) patient screening and written feedback of screening information to primary care clinicians, 3) clinician education on practice guidelines , 4) structured feedback between primary care and mental health clinicians, 5) continuity of patient care, and 6) a resource guide detailing available community services where the CHC has established reciprocal referrals. All of the intervention components will be implemented through the CM, except for the clinician education component, which will combine onsite and online continuing medical education (CME)-accredited sessions.
- Treatment-as-Usual (TAU): The TAU condition consists of only the clinician education and patient screening without written feedback.
Arm/Group | PTSD Care Management (PCM) | Treatment-as-Usual (TAU)
Serious Adverse Events (participants affected / at risk) | 0/206 | 0/198
Other Adverse Events (participants affected / at risk) | 20/206 | 23/198
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTSD Care Management (PCM) (N=206) | Treatment-as-Usual (TAU) (N=198)
suicidal ideation (Psychiatric disorders) | 20 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes